CLINICAL TRIAL: NCT01131520
Title: SBIRT in New Mexico
Brief Title: Screening Brief Intervention Referral to Treatment (SBIRT) in New Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-08-173; R01DA026003 (NIH)
Record Dates: First submitted 2010-05-21; First posted 2010-05-27 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Drug Abuse; HIV Risk Behavior
Keywords: SBIRT; Drug abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computerized Brief Intervention (Experimental): Computerized one-session brief intervention for drug use
  Interventions: Behavioral: Computerized brief intervention
- Counselor delivered brief intervention (Active Comparator): This is a brief intervention focused on drug use delivered by a behavioral health counselor and based on motivational interviewing
  Interventions: Behavioral: Counselor delivered brief intervention

INTERVENTIONS:
Behavioral: Computerized brief intervention — This is a brief computerized intervention focused on drug use of patients receiving primary care treatment in an outpatient setting. The intervention is delivered in one session.
  Arms: Computerized Brief Intervention
Behavioral: Counselor delivered brief intervention — This is a one session brief intervention delivered in a primary care setting that is based on motivational interviewing.
  Arms: Counselor delivered brief intervention

SUMMARY:
The purpose of this study is to compare the effectiveness in reducing drug use and its associated problems of a brief intervention for drug use delivered by a behavioral health counselor as compared to a brief intervention delivered by a computerized intervention.

DETAILED DESCRIPTION:
Drug use is a significant cause of morbidity and mortality in the United States. Efforts to develop and rigorously evaluate methods to provide Screening, Brief Intervention and Referral to Treatment (SBIRT) for drug users are needed. Computerized screening and brief interventions in particular have the potential to circumvent some of the potential problems of integrating SBIRT delivered by a counselor into busy primary care settings. These interventions may reduce drug use among individuals who are using drugs but are not yet drug dependent.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Moderate risk category on the ASSIST scores

Exclusion Criteria:

* planning to move out of New Mexico in the next year
* receipt of formal drug abuse treatment or a brief intervention for drug use in the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Schwartz, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Gryczynski J, Carswell SB, O'Grady KE, Mitchell SG, Schwartz RP. Gender and ethnic differences in primary care patients' response to computerized vs. in-person brief intervention for illicit drug misuse. J Subst Abuse Treat. 2018 Jan;84:50-56. doi: 10.1016/j.jsat.2017.10.009. Epub 2017 Nov 7. PMID 29195593
- [Derived] Mitchell SG, Monico LB, Gryczynski J, O'Grady KE, Schwartz RP. Staff Views of Acceptability and Appropriateness of a Computer-Delivered Brief Intervention for Moderate Drug and Alcohol Use. J Psychoactive Drugs. 2015 Sep-Oct;47(4):301-7. doi: 10.1080/02791072.2015.1075631. Epub 2015 Sep 16. PMID 26375411
- [Derived] Gryczynski J, Mitchell SG, Ondersma SJ, O'Grady KE, Schwartz RP. Potential radiating effects of misusing substances among medical patients receiving brief intervention. J Subst Abuse Treat. 2015 Aug;55:39-44. doi: 10.1016/j.jsat.2015.02.003. Epub 2015 Feb 23. PMID 25812927
- [Derived] Gryczynski J, Mitchell SG, Gonzales A, Moseley A, Peterson TR, Ondersma SJ, O'Grady KE, Schwartz RP. A randomized trial of computerized vs. in-person brief intervention for illicit drug use in primary care: outcomes through 12 months. J Subst Abuse Treat. 2015 Mar;50:3-10. doi: 10.1016/j.jsat.2014.09.002. Epub 2014 Sep 16. PMID 25282578
- [Derived] Schwartz RP, Gryczynski J, Mitchell SG, Gonzales A, Moseley A, Peterson TR, Ondersma SJ, O'Grady KE. Computerized versus in-person brief intervention for drug misuse: a randomized clinical trial. Addiction. 2014 Jul;109(7):1091-8. doi: 10.1111/add.12502. Epub 2014 Mar 10. PMID 24520906

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Started | 180 | 180
Completed | 179 | 176
Not Completed | 1 | 4
Not completed — Computer problem | 1 | 0
Not completed — Counselor not available | 0 | 3
Not completed — Subject changed history after enrollment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention | Total
Number analyzed (Participants) | 180 | 179 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (14.7) | 35.7 (14.6) | 36.1 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 82 | 165
  Male | 97 | 97 | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 85 | 168
  Not Hispanic or Latino | 97 | 94 | 191
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 12
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 3 | 1 | 4
  White | 162 | 161 | 323
  More than one race | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 180 | 179 | 359

OUTCOME MEASURES:

1. Primary Outcome: Alcohol, Smoking & Substance Involvement Screening Test (ASSIST) Score
Description: The ASSIST's Global Continuum of Illicit Drug Risk was used. A higher score is considered more severe risk. The scores range from 0 to 308.
Time Frame: 3 months post-baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Number analyzed (Participants) | 180 | 179
units on a scale | 27.8 (0.93) | 29.6 (0.93)

2. Primary Outcome: Hair Testing
Description: The number of participants testing positive on Radioimmunoassay (RIA) Hair Testing for opiates, cocaine, amphetamine and tetrahydrocannabinol (THC)
Time Frame: 3 month post-baseline
Population: The number of participants of the total sample who agreed to provide an analyzable hair specimen. Hair testing was not available for subjects not interviewed, those who refused testing, or who were unable to provide a sufficient quantity of hair for testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Number analyzed (Participants) | 159 | 155
Participants | 93 | 100

3. Secondary Outcome: Human Immunodeficiency Virus (HIV) Drug Use Risk Assessment Battery Subscale
Description: HIV Drug Use Risk Assessment Battery Subscale Score ranges from 0 to 22. A higher score is considered to be associated with higher risk.
Time Frame: 3 months post-baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Number analyzed (Participants) | 180 | 179
units on a scale | .06 (.03) | .01 (.03)

4. Secondary Outcome: Alcohol, Smoking & Substance Involvement Screening Test (ASSIST) Score
Description: ASSIST's Global Continuum of Illicit Drug Risk Score which ranges from 0 to 308. A higher score is associated with higher risk.
Time Frame: 6 month post-baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Number analyzed (Participants) | 180 | 179
units on a scale | 27.3 (1.30) | 27.4 (1.33)

5. Secondary Outcome: Alcohol, Smoking & Substance Involvement Screening Test (ASSIST) Score
Description: as for outcome 4
Time Frame: 12 months post-baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Number analyzed (Participants) | 180 | 179
units on a scale | 26.5 (1.32) | 25.9 (1.34)

6. Secondary Outcome: Hair Testing
Description: The predicted probabilities for testing positive on Radioimmunoassay (RIA) Hair Testing for opiates, cocaine, amphetamine and tetrahydrocannabinol (THC), calculated from generalized estimating equations.
Time Frame: 6 month post-baseline
Population: The sample includes participants who provided usable hair testing data at baseline.
Measure: Least Squares Mean (Standard Error); unit: predicted probability of positive test
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Number analyzed (Participants) | 159 | 155
predicted probability of positive test | .59 (.04) | .67 (.04)

7. Secondary Outcome: Hair Testing
Description: Predicted Probabilities for testing positive on the Radioimmunoassay (RIA) Hair Testing for opiates, cocaine, amphetamine and THC, calculated from generalized estimating equations.
Time Frame: 12 month post-baseline
Population: The sample includes participants who provided usable hair testing data at baseline
Measure: Least Squares Mean (Standard Error); unit: predicted probability of positive test
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Number analyzed (Participants) | 159 | 155
predicted probability of positive test | .57 (.04) | .59 (.04)

8. Secondary Outcome: Human Immunodeficiency Virus (HIV) Risk Assessment Battery Subscale
Description: as for outcome 3
Time Frame: 6 month post-baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Number analyzed (Participants) | 180 | 179
units on a scale | .02 (.03) | .04 (.03)

9. Secondary Outcome: Human Immunodeficiency Virus (HIV) Risk Assessment Battery Subscale Score
Description: as for outcome 3
Time Frame: 12 month post-baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Number analyzed (Participants) | 180 | 179
units on a scale | .05 (.03) | .01 (.04)

ADVERSE EVENTS:
Arm/Group | Computerized Brief Intervention | Counselor Delivered Brief Intervention
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/179
Other Adverse Events (participants affected / at risk) | 0/180 | 0/179

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes